CLINICAL TRIAL: NCT00611715
Title: A Phase II Trial of Letrozole Plus OSI-774 (Tarceva) in Post-menopausal Women With ER and/or PR-Positive Metastatic Breast Cancer
Brief Title: Ph II Letrozole + OSI-774 (Tarceva) in Post-menopausal, w/ ER and/or PR-positive Met Breast Cancer.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ingrid Mayer, MD, Assistant Professor of Medicine; Clinical Director, Breast Cancer Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 0303; VU-VICC-BRE-0303; VU-VICC-030592; GENENTECH-VU-VICC-BRE-0303; NOVARTIS-VU-VICC-BRE-0303; NCT00179296 (obsolete NCT alias)
Record Dates: First submitted 2008-02-08; First posted 2008-02-11 (Estimated); Results first posted 2012-07-13 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Erlotinib Hydrochloride; Letrozole; In Situ Hybridization, Fluorescence; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- First line/hormone-therapy naive (Experimental)
  Interventions: Drug: erlotinib hydrochloride; Drug: letrozole; Genetic: fluorescence in situ hybridization; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis
- Second-line/prev hormone-therapy tx (Experimental)
  Interventions: Drug: erlotinib hydrochloride; Drug: letrozole; Genetic: fluorescence in situ hybridization; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — OSI-774 150 mg/day
  Other Names: Tarceva, OSI-774
Drug: letrozole — Letrozole 2.5 mg/day
  Other Names: Femara
Genetic: fluorescence in situ hybridization — To determine HER2 gene amplification or excess copies of the HER2 gene
  Other Names: None specified
Other: immunohistochemistry staining method — to measure the epidermal growth factor receptors (EGFR)
  Other Names: None specified
Other: laboratory biomarker analysis — To determine if specific biomarkers exhibit a longer time to tumor progression after treatment with the study drugs
  Other Names: none specified

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by blocking the use of estrogen by the tumor cells. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving letrozole together with erlotinib may kill more tumor cells.

PURPOSE: This phase II clinical trial is studying how well giving letrozole together with erlotinib works in treating postmenopausal women with estrogen receptor-positive and/or progesterone receptor-positive locally recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the rate of clinical benefit (complete response [CR], partial response [PR], and stable disease [SD] in patients with hormone-dependent locally recurrent or metastatic breast cancer treated with letrozole in combination with erlotinib hydrochloride.

Secondary

* To determine the time to progression (TTP) in patients treated with this regimen.
* To evaluate the anti-tumor activity, as determined by CR and PR rates, of this regimen in these patients.
* To evaluate the safety of this regimen in these patients.
* To determine if tumors that are positive for epidermal growth factor receptor (EGFR) or Ser118 ER, or that overexpress human epidermal receptor (HER2) exhibit a longer TTP from the combination compared to tumors that do not express or overexpress these molecules.

OUTLINE: This is a multicenter study. Patients are stratified according to prior hormone therapy (hormone-therapy naive/first-line therapy vs prior hormonal therapy with either tamoxifen or an aromatase inhibitor in the adjuvant or metastatic setting/second-line therapy)

Patients receive oral letrozole and oral erlotinib hydrochloride once daily in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then yearly thereafter.

ELIGIBILITY:
* Patients must have estrogen (ER) and/or progesterone receptor (PgR)-positive, histologically confirmed adenocarcinoma of the breast with measurable (but not operable) locally recurrent disease, or measurable and/or evaluable metastatic disease (see protocol section 10.3), including isolated bone metastases.
* Patients with available paraffin tissue blocks from either the primary or the metastatic site must submit tissue blocks for retrospective EGFR and HER2 analysis. If tissue blocks cannot be submitted, 20 unstained slides from each paraffin block must be submitted.
* All patients must be post-menopausal females as defined by one of the following:

  * Prior bilateral oophorectomy
  * Prior bilateral ovarian irradiation
  * No menstrual period for 12 months or longer
  * If age 55 years or less and < 12 months from last menstrual period, patient must have a serum estradiol < or equal to 30 and an FSH level > 40.
* Patients must not have had more than 1 prior chemotherapy regimen for metastatic disease and have fully recovered from any grade 2-4 toxicities related to chemotherapy. No concurrent chemotherapy is allowed while on protocol therapy.
* Patients may have had 1 prior hormonal therapy for metastatic disease. This includes: tamoxifen, fulvestrant, anastrozole, exemestane, aminoglutethimide, megace, and letrozole. Patients may have received tamoxifen or aromatase inhibitors in the adjuvant setting.
* Patients must not have had prior therapy with EGF receptor inhibitors.
* Previous but not concomitant therapy with trastuzumab (Herceptin) is allowed. Patients must not have received Herceptin within 4 weeks of initiation of protocol therapy.
* Patients must have an ECOG performance status of 0, 1, or 2.
* Patients must have adequate hematologic, hepatic, and renal function as defined by the following within 2 weeks of initiation of therapy:

  * Absolute neutrophils > or equal to 1,500/mm3 and platelets > or equal to 100,000/mm3.
  * Bilirubin < than or equal to 1.5 upper limit of normal.
  * SGOT and SGPT < or equal to 2.5 upper limit of normal.
  * Creatinine < or equal to 1.5 upper limit of normal.
  * INR, PTT and PT in the normal range.
  * Must be 18 years of age or older.
* Patients must not have a history of central nervous system metastases or unevaluated CNS symptoms suggestive of possible brain metastases.
* Patients may receive concurrent radiation therapy to painful bone metastases or areas of impending bone fracture as long as radiation therapy is initiated prior to study entry and sites of evaluable disease outside the radiation port(s) are available for follow-up. Patients who have received prior radiotherapy must have recovered from toxicity induced by this treatment.
* Patients < 55 years of age must not have received Luteinizing hormone releasing hormone (LHRH) antagonists within 3 months prior to protocol therapy.
* Patients must not suffer from medical or psychiatric conditions that would interfere with ability to provide informed consent, communicate side effects, or comply with protocol requirements including maintenance of a compliance/pill diary.
* Patients must be disease-free of prior invasive cancers for > 5 years with the exception of basal or squamous cancer of the skin or cervical carcinoma in situ.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2003-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mayer, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (9):
- United States (9):
  - Central Georgia Hematology/Oncology Associates, P.C., Macon, Georgia
  - Jennie Stuart Medical Center, Hopkinsville, Kentucky
  - Purchase Cancer Group, Paducah, Kentucky
  - Memorial Health Care System, Chattanooga, Tennessee
  - The Jones Clinic - Germantown, Germantown, Tennessee
  - Jackson-Madison County Hospital, Jackson, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients from November 2003 through July 2008.
Pre-assignment Details: Fifty-one patients consented, one was ineligible and two withdrew before receiving study drug.
Groups:
- First Line/Hormone-therapy Naive: Patients who have not received hormonal therapy
- Second-line/Prev Hormone-therapy tx: Patients who have previously received hormonal therapy
Period: Overall Study
Arm/Group | First Line/Hormone-therapy Naive | Second-line/Prev Hormone-therapy tx
Started | 42 | 6
Completed | 1 (2 pts in Arm 1 remain on-tx. They are not accounted for in "off-tx reason"or "completed" data fields) | 0
Not Completed | 41 | 6
Not completed — Disease Progression | 24 | 4
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Adverse Event | 9 | 1
Not completed — Death | 1 | 0
Not completed — two patients are still on treatment | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Line/Hormone-therapy Naive | Second-line/Prev Hormone-therapy tx | Total
Number analyzed (Participants) | 42 | 6 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 5 | 29
  >=65 years | 18 | 1 | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (1) | 54 (1) | 61 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 6 | 48
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 6 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pathological Complete Response.
Description: Per RECIST criteria v. 1.0: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions
Time Frame: at 24 weeks
Population: Analysis population is patients who were available for response measurement. Some patients did not meet the criteria to be analyzed for response evaluation which accounts for the discrepancy in patients analyzed vs. total accrual population.
Measure: Number; unit: participants
Groups:
- Hormone Therapy Naive: Patients who were endocrine treatment-naïve in the metastatic setting and more than 12 months from adjuvant endocrine therapy. They received Letrozole 2.5 mg/day and OSI-774 150 mg/day, both orally.
- Previous Hormone Therapy: Patients who had either received one line of endocrine therapy in the metastatic setting or recurred less than 12 months after completion of endocrine therapy. They received Letrozole 2.5 mg/day and OSI-774 150 mg/day, both orally.
Arm/Group | Hormone Therapy Naive | Previous Hormone Therapy
Number analyzed (Participants) | 35 | 5
participants | 28 | 0

2. Secondary Outcome: Median Time to Progression of Target Lesions
Description: Time frame from study entry till discontinuation of treatment due to disease progression. Progression of target lesions is measured by RECIST criteria v. 1.0: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, progressive disease (PD) > 20% increase in the sum of the LD of target lesions or appearance of new lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions.
Time Frame: Every 12 weeks from on-study to disease progression
Population: Patients who were available for response measurement. Seven patients in the Hormone therapy naive arm did not meet the criteria for response evaluation. One patient in the Previous Hormone Therapy arm did not meet the criteria for response evaluation.
Measure: Median (Full Range); unit: Months
Groups:
- First Line/Hormone-therapy Naive: Patients who were endocrine treatment-naïve in the metastatic setting and more than 12 months from adjuvant endocrine therapy. They received Letrozole 2.5 mg/day and OSI-774 150 mg/day, both orally.
- Second-line/Prev Hormone-therapy tx: Patients who had either received one line of endocrine therapy in the metastatic setting or recurred less than 12 months after completion of endocrine therapy. They received Letrozole 2.5 mg/day and OSI-774 150 mg/day, both orally.
Arm/Group | First Line/Hormone-therapy Naive | Second-line/Prev Hormone-therapy tx
Number analyzed (Participants) | 35 | 5
Months | 12 (11.5) [1 to 75] | 3 (0) [2 to 4]

3. Secondary Outcome: Number of Patients With Anti-tumor Activity: Complete Response (CR) and Partial Response (PR)
Description: Per RECIST criteria v. 1.0: measurable lesions: complete response (CR) disappearance of target lesions and partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions.
Time Frame: at 24 weeks
Population: Analysis population is patients who were available for response measurement. Seven patients in the Hormone therapy naive arm did not meet the criteria for response evaluation. One patient in the Previous Hormone Therapy arm did not meet the criteria for response evaluation.
Measure: Number; unit: participants
Groups:
- First Line/Hormone-therapy Naive: Patients that were endocrine treatment-naive in the metastatic setting and more than 12 months from adjuvant endocrine therapy
- Second-line/Prev Hormone-therapy tx: Patients that had either received one line of endocrine therapy in the metastatic setting or recurred less than 12 months after completion of endocrine therapy
Arm/Group | First Line/Hormone-therapy Naive | Second-line/Prev Hormone-therapy tx
Number analyzed (Participants) | 35 | 5
participants | 8 | 0

4. Secondary Outcome: Number of Patients With Worst-grade Toxicities Per Grade
Description: Number of patients with worst-grade toxicities following NCI Common Toxicity Criteria: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, disabling, 5 = death
Time Frame: at 24 weeks
Population: All patients who received treatment and experienced an adverse event.
Measure: Number; unit: participants
Groups:
- First Line/Hormone-therapy Naive: Patients that were endocrine treatment-naïve in the metastatic setting and more than 12 months from adjuvant endocrine therapy. They received Letrozole 2.5 mg/day and OSI-774 150 mg/day, both orally.
- Second-line/Prev Hormone-therapy tx: Patients that had either received one line of endocrine therapy in the metastatic setting or recurred less than 12 months after completion of endocrine therapy. They received Letrozole 2.5 mg/day and OSI-774 150 mg/day, both orally.
Arm/Group | First Line/Hormone-therapy Naive | Second-line/Prev Hormone-therapy tx
Number analyzed (Participants) | 42 | 6
participants
  Worst grade toxicity Grade 1 | 11 | 0
  Worst grade toxicity Grade 2 | 21 | 3
  Worst grade toxicity Grade 3 | 8 | 2
  Worst grade toxicity Grade 4 | 1 | 0
  Worst grade toxicity Grade 5 | 0 | 0

ADVERSE EVENTS:
Arm/Group | First Line/Hormone-therapy Naive | Second-line/Prev Hormone-therapy tx
Serious Adverse Events (participants affected / at risk) | 20/42 | 1/6
Other Adverse Events (participants affected / at risk) | 2/42 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Line/Hormone-therapy Naive (N=42) | Second-line/Prev Hormone-therapy tx (N=6)
catheter-related infection (Infections and infestations) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 3 (4) | 0 (0)
creatinine (Investigations) | 1 (1) | 0 (0)
cellulitis, breast (Infections and infestations) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0)
cebebrovascular ischema (Vascular disorders) | 1 (1) | 0 (0)
infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0)
acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
alkaline phosphate (Investigations) | 1 (1) | 0 (0)
bilirubin (Investigations) | 1 (1) | 0 (0)
transaminases elevation (Investigations) | 2 (4) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (4) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
thrombosis (Vascular disorders) | 1 (1) | 0 (0)
infection - urinary (Infections and infestations) | 1 (1) | 0 (0)
neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
pericardial effusion (Cardiac disorders) | 1 (2) | 0 (0)
hypotension (Vascular disorders) | 1 (1) | 0 (0)
hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
death (General disorders) | 2 (2) | 0 (0)
arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
platelets (Investigations) | 1 (1) | 0 (0)
edema (General disorders) | 1 (1) | 0 (0)
pain, breast (General disorders) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 2 (8) | 0 (0)
hot flash (Vascular disorders) | 1 (1) | 0 (0)
anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
headache (Nervous system disorders) | 3 (3) | 0 (0)
creatinine (Investigations) | 2 (3) | 0 (0)
hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
fatigue (General disorders) | 1 (2) | 0 (0)
confusion (Psychiatric disorders) | 1 (1) | 0 (0)
joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
sinus tachycardia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Blood urea nitrogen (BUN) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
fever (General disorders) | 1 (1) | 1 (5)
keratitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Line/Hormone-therapy Naive (N=42) | Second-line/Prev Hormone-therapy tx (N=6)
hemoglobin increased (Investigations) | 2 (7) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0)
skin rash (Skin and subcutaneous tissue disorders) | 2 (8) | 0 (0)
insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
hypertension (Vascular disorders) | 2 (2) | 0 (0)
neuropathy (Nervous system disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The total number of worst-grade toxicities will not match the total number of participants, as patients can have multiple events or no events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes